CLINICAL TRIAL: NCT02963987
Title: Effect of Portion Size Over 5 Days in Preschool Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); United States Department of Agriculture (USDA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Barbara J. Rolls, Professor of Nutrition and Director of the Laboratory for the Study of Human Ingestive Behavior, Penn State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: ChildFood501; R01DK082580 (NIH); 2011-67001-30117 (Other Grant/Funding Number: United States Department of Agriculture)
Record Dates: First submitted 2016-11-10; First posted 2016-11-15 (Estimated); Results first posted 2019-05-29 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-05

CONDITIONS: Feeding Behavior
MeSH Terms: conditions — Feeding Behavior | interventions — Food

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 100% Portion Size (Experimental): 100% Food and Beverage Portion Size
  Interventions: Other: Food and Beverage Portion Size
- 150% Portion Size (Experimental): 150% Food and Beverage Portion Size
  Interventions: Other: Food and Beverage Portion Size

INTERVENTIONS:
Other: Food and Beverage Portion Size — Variations of Food and Beverage Portion Size (100% Baseline portions and increased 50% for 150% portions)

SUMMARY:
In this study, the investigators varied the portion size of all meals served during two 5-day periods. During one period, baseline amounts of all foods and beverages were served, and during the other, the portion size of all items was increased by 50%. The primary aim of the study is to determine the effect of varying the portion size of foods and beverages served over 5 days on energy intake in preschool children.

ELIGIBILITY:
Inclusion Criteria:

* Attending one of the designated childcare centers

Exclusion Criteria:

* Food Allergies
* Food Restrictions
* Health Issues that Preclude Participation
* Not available for duration of the study

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Laboratory for the Study of Human Ingestive Behavior, University Park, Pennsylvania
  - The Pennsylvania State University, Laboratory for the Study of Human Ingestive Behavior, University Park, Pennsylvania

REFERENCES:
- [Result] Smethers AD, Roe LS, Sanchez CE, Zuraikat FM, Keller KL, Kling SMR, Rolls BJ. Portion size has sustained effects over 5 days in preschool children: a randomized trial. Am J Clin Nutr. 2019 May 1;109(5):1361-1372. doi: 10.1093/ajcn/nqy383. PMID 30976782
- [Derived] Roe LS, Keller KL, Rolls BJ. Food Properties and Individual Characteristics Influence Children's Intake Across Multiple Days of Weighed Assessments in Childcare Programs. J Nutr. 2023 May;153(5):1646-1655. doi: 10.1016/j.tjnut.2023.03.025. Epub 2023 Mar 24. PMID 36965692

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants for the study were recruited from 7 classrooms of 2 childcare centers in University Park, PA from June 2015 to April 2016.
Groups:
- 100% Portion Size First, Then 150% Portion Size: 100% Food and Beverage Portion Size in first period, then 150% Food and Beverage Portion Size in second period
- 150% Portion Size First, Then 100% Portion Size: 150% Food and Beverage Portion Size in first period, then 100% Food and Beverage Portion Size in second period
Period: First Intervention Period
Arm/Group | 100% Portion Size First, Then 150% Portion Size | 150% Portion Size First, Then 100% Portion Size
Started | 31 | 19
Completed | 31 | 19
Not Completed | 0 | 0
Period: Second Intervention Period
Arm/Group | 100% Portion Size First, Then 150% Portion Size | 150% Portion Size First, Then 100% Portion Size
Started | 31 | 19
Completed | 31 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Data of 4 enrolled participants was excluded from analysis for absence from meals on 3 or more days in one intervention period
Groups:
- All Study Participants: All participants in the crossover trial of two interventions in two periods
Arm/Group | All Study Participants
Number analyzed (Participants) | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.3 (0.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 35
  Unknown or Not Reported | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 34
  More than one race | 3
  Unknown or Not Reported | 5
Region of Enrollment [Number; unit: participants]
  United States | 46

OUTCOME MEASURES:

1. Primary Outcome: Differences in Food and Beverage Intake by Energy
Description: Differences between 100% and 150% portion size conditions in energy intake (kcal) determined from weighed intakes of food and beverages
Time Frame: Days 1-5 in Periods 1 and 2
Population: as for baseline characteristics
Measure: Mean (Standard Error); unit: kilocalories
Groups:
- 100% Portion Size: 100% Food and Beverage Portion Size (baseline portions)
- 150% Portion Size: 150% Food and Beverage Portion Size (increased 50% from baseline portions)
Arm/Group | 100% Portion Size | 150% Portion Size
Number analyzed (Participants) | 46 | 46
kilocalories | 914 (44) | 1081 (44)
Statistical Analysis 1: Comparison: 100% Portion Size vs 150% Portion Size; Test type: Superiority; p < 0.0001, Mixed Models Analysis

2. Secondary Outcome: Differences in Food and Beverage Intake by Energy Density
Description: Differences between 100% and 150% portion size conditions in daily energy density (kcal/g) determined from weighed intakes of food and beverages
Time Frame: Days 1-5 in Periods 1 and 2
Population: as for baseline characteristics
Measure: Mean (Standard Error); unit: kilocalories/gram
Groups:
- 100% Portion Size: 100% Food and Beverage Portion Size
  Food and Beverage Portion Size: Variations of Food and Beverage Portion Size, 100% Baseline portions and increased 50% for 150% portions
- 150% Portion Size: 150% Food and Beverage Portion Size
  Food and Beverage Portion Size: Variations of Food and Beverage Portion Size, 100% Baseline portions and increased 50% for 150% portions
Arm/Group | 100% Portion Size | 150% Portion Size
Number analyzed (Participants) | 46 | 46
kilocalories/gram | 1.45 (0.04) | 1.50 (0.04)
Statistical Analysis 1: Comparison: 100% Portion Size vs 150% Portion Size; Test type: Superiority; p = 0.006, Mixed Models Analysis

3. Secondary Outcome: Differences in Food and Beverage Intake by Weight
Description: Differences between 100% and 150% portion size conditions in daily weighed intake of food and beverages (g)
Time Frame: Days 1-5 in Periods 1 and 2
Population: as for baseline characteristics
Measure: Mean (Standard Error); unit: grams
Arm/Group | 100% Portion Size | 150% Portion Size
Number analyzed (Participants) | 46 | 46
grams | 899 (45) | 1042 (46)
Statistical Analysis 1: Comparison: 100% Portion Size vs 150% Portion Size; Test type: Superiority; p < 0.0001, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 5 weeks
Groups:
- 100% Portion Size: Study participants in the period in which they were served 100% portions of food and beverages. The total includes participants who were served some meals but whose data was excluded from analysis for low attendance.
- 150% Portion Size: Study participants in the period in which they were served 150% portions of food and beverages. The total includes participants who were served some meals but whose data was excluded from analysis for low attendance.
Arm/Group | 100% Portion Size | 150% Portion Size
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No